CLINICAL TRIAL: NCT06574529
Title: Video-observed Therapy (vDOT) as a Surrogate to Directly Observed Therapy (DOT) for Active Tuberculosis: a Feasibility Study in a Low Incidence High-income Area
Brief Title: Video-observed Therapy for Active Tuberculosis: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ligue Pulmonaire Genevoise (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCER 2021-01713
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis Active
Keywords: Compliance; Directly observed therapy; Video-observed therapy
MeSH Terms: conditions — Tuberculosis; Patient Compliance; Directly Observed Therapy

STUDY DESIGN:
Intervention Model Description: All patients with active tuberculosis were invited to participate in the study and followed during the duration of their treatment until treatment completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): The study is not randomised; all subjects included are submitted to the VOT
  Interventions: Device: Video-observed therapy (vDOT)

INTERVENTIONS:
Device: Video-observed therapy (vDOT) — All participants are required to send 5 times per week a short video showing they are actually taking their treatment for tuberculosis via a dedicated application on their cellphone

SUMMARY:
Tuberculosis (TB) is still present in Switzerland, and concerns mainly foreign-born subjects. Monitoring compliance to treatment by Directly Observed Therapy (DOT) is strongly encouraged by the World Health Organization (WHO). It is however time-consuming, costly and stigmatising. This study aims to examine the feasibility of monitoring compliance through a secured web platform and videos sent via an application on a cellphone, a concept known as vDOT (Video-observed therapy). The study aims to include all patients treated for tuberculosis is on our area during an 18 month period and monitor acceptance, compliance, and technical issues related to vDOT.

DETAILED DESCRIPTION:
The study aims to include all patients who are treated de novo for active tuberculosis is our area. The aim of this study, was to show that vDOT was feasible in a low-incidence high income area, that it had a high acceptance rate among patients and health-care professionals, with a low rate of technical difficulties or pitfalls.

All patients with a diagnosis of tuberculosis irrespective of site(s) of infection, were invited to participate in this study. The Division of Pulmonology of Geneva University Hospital diagnoses and follows virtually all cases of tuberculosis in the Canton of Geneva. Annual number of cases in Geneva between 2020 and 2023 was on average 43/year (range: 36-53). Incidence was 7-10.3/105 inhabitants compared to a national incidence of 3.99-4.72 /105 inhabitants during the same period.

Specialized TB nurses were trained to use the vDOT platform and provided the training with the help of translators whenever required. The application (APP) was installed with the patient, and a test video was sent to the platform. The APP uses simple understandable pictograms and is thus not per se language-dependent . vDOT was started as soon as possible after initiation of TB treatment, either during a hospital stay or during the first outpatient follow-up visit at our centre. Whenever necessary, a portable cell phone was provided for the patient, for the duration of the treatment.

The SureAdhere platform was used for vDOT (https://dimagi.com/sureadhere/). Once the videos have been recorded, they are sent automatically as soon as the patients' cell phone has access to internet.

For each patient, the number of videos to be sent each week was specified (5 as default option).

ELIGIBILITY:
Inclusion Criteria:

* age above 16 years of age; providing informed consent (translators were used whenever necessary to ensure understanding of study and vDOT procedure); having a diagnosis of untreated active tuberculosis, irrespective of site of infection, confirmed by culture and/or Polymerase chain reaction test (PCR) and follow-up ensured by Geneva University Hospital.

Exclusion Criteria:

* refusal to participate, not fulfilling inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Acceptance rate | Two weeks after starting TB treatment
  Number of patients accepting to install the application on their cellphone and send videos of their treatment until treatment completion, among all patients initiating a treatment for active tuberculosis in our center
Effective implementation rate | Two weeks after starting TB treatment
  Number of patients for whom installing the application, and learning how to use it was possible among all patients with active TB during study period

SECONDARY OUTCOMES:
Ratio of number of videos sent to number of videos expected | Duration of treatment (max 12 months)
  Number of videos recorded on the secured platform compared with number expected(% x number of weeks of treatment)
Quality of videos sent | Duration of treatment (max 12 months)
  Proportion of videos with technical problems (sound, lighting, framing) was recorded
Evaluation of video-observed therapy by specialized nurses following the patients | End of study (18 months)
  Questionnaire with Likert scales submitted to all nurses at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No